CLINICAL TRIAL: NCT05421936
Title: Uncommon EGFR Mutations: International Case Series on Efficacy of Osimertinib in Real-life Practice in First Line Setting
Brief Title: Osimertinib for NSCLC With Uncommon EGFR Mutations
Acronym: UNICORN
Status: Suspended | Type: Observational
Why Stopped: Result summarized and published
Sponsor: Sheba Medical Center (Other Government)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Jair Bar, M.D., Ph.D., Head of Thoracic Oncology Unit, Institute of Oncology, Sheba Medical Center
Other Study IDs: UNICORN_226_13
Record Dates: First submitted 2022-03-30; First posted 2022-06-16 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Genes, erbB-1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Osimertinib — Treatment as the first EGFR-TKI

SUMMARY:
This is a multi-center, retrospective study of ucEGFRmut (exon 20 insertions excluded) metastatic NSCLC osimertinib-treated as first EGFR inhibitor. RECIST and RANO-BM brain objective response rate (ORR) were evaluated by investigators. mPFS, mOS and mDOR were calculated from osimertinib initiation. Mutations found at resistance were collected.

DETAILED DESCRIPTION:
The epidermal growth factor receptor ( EGFR) is the most common targetable driver in non-small cell lung cancer (NSCLC). Approximately 90% of the EGFR mutations include an exon 19 deletion and a L858R point mutation at exon 21. Less common mutations include, among others, G719X in exon 18, L861Q in exon 21, exon 20 insertions, S768I in exon 20, and T790M in exon 20. Osimertinib is an EGFR TKI that has been developed as non-competitive inhibitor targeting a range of EGFR mutant molecules, currently regarded as the first-line treatment of choice to EGFR mutant (EGFRm) patients. Inhibition of the less common EGFR mutant by osimertinib has been demonstrated.

Real-world data showed lower response rate (RR) and progression free survival (PFS) in patients harboring uncommon EGFR mutations compared to the ones with common mutations treated with EGFR TKIs. Osimertinib as treatment for patients with rare mutations has been assessed in a single arm phase II study in Korea. RR was 50%, PFS was 8.2 months, mOS was not reached. Osimertinib activity in patients with uncommon mutations was assessed also in a retrospective US study, time on treatment ranged from 7.7 months to 19.3 months.

This is a multi-centric, retrospective, real-world study. Study goal is to collect high quality data regarding the efficacy of osimertinib in TKI naive NSCLC patients with uncommon EGFR mutations. The primary endpoints are progression-free survival and overall survival, from osimertinib start. Secondary endpoints would be RECIST response, adverse events, time on treatment and time to CNS progression, CNS response and mechanisms of resistance if tested.

The study includes researchers from Belgium, Denmark, Israel, Switzerland, Netherlands, Germany, France, Italy and USA. Data collection will be conducted at each participating site, following ethics approval. No patient identifying information will leave each of the participating centers. Data will be collected centrally by the lead investigators and analyzed for the entire study cohort and for subgroups if deemed appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. NSCLC by histologic or cytologic diagnosis
3. Stage IV or stage III not amendable to curative treatment (i.e., advanced disease)
4. Uncommon mutation of EGFR (exon 20 insertion excluded)
5. Treated with osimertinib for advanced disease as first TKI
6. Osimertinib initiated not later than end of January 2021

Exclusion criteria:

1. Lack of any follow-up data
2. Lack of consent for data collection or ethics committee approval for the waiver of informed consent (i.e. for deceased patients)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced NSCLC with uncommon EGFR mutation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-27 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From date of osimertinib initiation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  investigator-defined PFS
Overall survival | From date of osimertinib initiation until date of death from any cause, assessed up to 100 months
  OS

SECONDARY OUTCOMES:
Overall response rate | From date of osimertinib initiation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  RECIST-defined ORR
Brain response | From date of osimertinib initiation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  RANO-BM
Adverse events on osimertinib | From date of osimertinib initiation until 30 days after the date of last osimertinib treatment or date of death from any cause, whichever came first, assessed up to 100 months
  Adverse events on osimertinib
Time on treatment (TOT, on osimertinib) | From date of osimertinib initiation until the date of last osimertinib treatment or date of death from any cause, whichever came first, assessed up to 100 months
  Time on treatment (TOT, on osimertinib)
Time to CNS progression | From date of osimertinib initiation until the date of first documented CNS progression or censured at last follow up or at date of death from any cause, whichever came first, assessed up to 100 months
  Time to CNS progression
Mechanisms of resistance | From date of osimertinib initiation until the date of molecular test performed after any documented progression, assessed up to 100 months
  Results of molecular tests done at time of progression on osimertinib (if done)

CONTACTS AND LOCATIONS:
Overall Officials: Jair Bar, MD-PhD, Principal Investigator — Sheba Medical Center, Ramat Gan, Israel; Alfredo Addeo, MD, Principal Investigator — Geneva University Hospital, Geneva, Switzerland
Locations (1):
- Sheba Medical Centre, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided